CLINICAL TRIAL: NCT02044549
Title: Carbetocin Versus Syntometrine for Prevention of Postpartum Hemorrhage After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Carbitocin
Record Dates: First submitted 2014-01-15; First posted 2014-01-24 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Postpartum Hemorrhage; Blood Loss
Keywords: Carbetocin; syntometrine; postpartum hemorrhage; cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — carbetocin; syntometrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- carbetocin (Active Comparator): single 100 μg IV dose of carbetocin (150 women) after fetal extraction and before placental removal.
  Interventions: Drug: carbetocin
- Syntometrine (Active Comparator): Intravenous combination of 5 IU oxytocin and 0.2 mg ergometrine (300 women) after fetal extraction and before placental removal.
  Interventions: Drug: Syntometrine

INTERVENTIONS:
Drug: carbetocin — Oxycontin analogue
  Other Names: Pabal
  Arms: carbetocin
Drug: Syntometrine — Uterotonins
  Other Names: Oxytocin methergine combination
  Arms: Syntometrine

SUMMARY:
to compare effectiveness and tolerability of carbetocin versus syntometrine in prevention of Postpartum hemorrhage after cesarean section

DETAILED DESCRIPTION:
A double blind randomized study conducted on 450 pregnant subjected randomly either to single 100 μg IV dose of carbetocin (150 women) or combination of 5 IU oxytocin and 0.2 mg ergometrine (300 women) after fetal extraction and before placental removal.

Prevention of postpartum haemorrhage (PPH) after cesarean section (CS) had been evaluated by measurement of drop of Hemoglobin and hematocrit, incidence of PPH and number of subjects needed additional oxytocic

ELIGIBILITY:
Inclusion Criteria:

* All participants are at 37 - 40 weeks of gestational age
* Noncomplicated pregnancy.

Exclusion Criteria:

* Participants with placenta previa
* Patients with coagulopathy
* preeclamptic women
* known sensitivity to oxytocin or methergine were excluded

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
prevention of post partum hemorrhage after CS | 24 hours
  Number of participants experienced postpartum hemorrhage

SECONDARY OUTCOMES:
side effects of drugs used | 24 hours
  Number of subjects experienced Hemodynamic changes (blood pressure , pulse and respiratory rate ) , GIT side effects as nausea , vomiting and metallic taste, Vasomotor effects as flushing, headache , itching

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Ass prof kasr aini medical school
Locations (1):
- Ahmed Maged, Cairo, Egypt